CLINICAL TRIAL: NCT05268718
Title: Gold-silver-cuprous Oxide (Au-Ag-Cu2O) Composite Nanogel Combined With Photothermal Therapy in the Treatment of Severe Drug-resistant Microbial Keratitis
Brief Title: Au-Ag-Cu2O NG With PTT Anti Drug-resistant Microbial Keratitis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0635
Record Dates: First submitted 2022-02-09; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2021-08

CONDITIONS: Keratitis, Ulcerative; Antibiotic Resistance, Microbial; Photothermal Therapy
Keywords: Photothermal Therapy; Keratitis, Ulcerative; Antibiotic Resistance, Microbial
MeSH Terms: conditions — Corneal Ulcer | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nanogel photothermal therapy (Experimental): After the subjects were enrolled in the study, the eyes were coated with Au-Ag-Cu2O nano-gel once (the concentration was 26.4μg/mL, the dosage was suitable to cover the ulcer surface evenly, and the dosage was recorded). Combined with mdl-n-808-10w near-infrared laser (China changchun new industry photoelectric technology) combined with photothermal therapy (laser wavelength 808 nm, power 1.5W/cm2, temperature controlled at 40℃, lasting 10min)
  Interventions: Drug: Hollow gold and silver alloy cuprous oxide shell nano-shell hydrogel
- Voriconazole eye drops (Active Comparator): Voliconazole eye drops (once in half an hour) were also used in the control group.
  Interventions: Drug: Voriconazole eye drops
- Normal saline (Placebo Comparator): Normal saline eye drops (once in half an hour) were also used in the control group.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Hollow gold and silver alloy cuprous oxide shell nano-shell hydrogel — Hollow gold and silver alloy cuprous oxide shell nano-shell hydrogel was excited by NIR laser to release functional silver ions, copper ions and ROS.
  Other Names: Au-Ag-Cu2O nano-gel
  Arms: Nanogel photothermal therapy
Drug: Voriconazole eye drops — Voriconazole eye drops (1%) were administrated to infectious eye very frequently (once half an hour)
  Other Names: VRC
  Arms: Voriconazole eye drops
Other: Normal saline — To be placebo, normal saline were administrated to infectious eye
  Other Names: NS
  Arms: Normal saline

SUMMARY:
This clinical study was conducted to evaluate the efficacy and safety of gold-silver cuprous oxide composite nanogels combined with photothermal therapy system in the treatment of severe drug-resistant bacterial keratitis ineffective by traditional antibiotic treatment in human eyes, and to provide translational applications. Based on the clinical evidence, a more effective and safe innovative treatment plan for corneal diseases has been developed.

ELIGIBILITY:
Inclusion Criteria:

1. The monocular cases of severe infectious keratitis admitted to our center were diagnosed as fungal keratitis according to their medical history, physical signs and surface secretions smear examination of corneal ulcer lesions (severe was defined as subjects with visual acuity < 0.15, deep stromal infiltration or involvement diameter >2mm, with extensive infiltration around or with extensive suppuration)
2. After more than 2 weeks of active treatment with antibiotics, there was no effect
3. The researchers communicated with the subjects in detail, and the subjects cooperated well and they voluntarily participated and signed informed consent

Exclusion Criteria:

1. Allergic to the drug in this test.
2. Pregnant and lactating women.
3. The medical history suggests serious heart, lung, liver, kidney dysfunction.
4. Patients with other factors that would affect the results of this result.
5. No signed informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Anterior segment photography | 1 month
  corneal edema, keratohelcosis, hppopyon
confocal microscopy | 1 month
  fungal hyphae in corneal surface

SECONDARY OUTCOMES:
eye pressure | 1 month
  Measurement of contact tonometry with iCare TA01i tonometer after treatment (1 day, 1 week, 1 month)
visual acuity | 1 month
  Measurement of distance visual acuity with subjective refraction after treatment (1 week, 1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Ke Yao, MD, Study Director — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China